CLINICAL TRIAL: NCT02908737
Title: Clinical Evaluation of Bass and Treble Controls for CI Subjects
Acronym: CLASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5640
Record Dates: First submitted 2016-08-19; First posted 2016-09-21 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bass and Treble controls (Experimental): Bass and Treble controls are clinician enabled and provide the recipient with access to the adjustment of low and high frequency sound balance, known as Bass and Treble respectively.
  Interventions: Device: Bass and Treble

INTERVENTIONS:
Device: Bass and Treble — Bass and Treble controls are clinician enabled and provide the recipient with access to the adjustment of low and high frequency sound balance, known as Bass and Treble respectively

SUMMARY:
The clinical study is designed to evaluate the safety and effectiveness of recipient controlled Bass and Treble.

DETAILED DESCRIPTION:
Bass and Treble controls provide the CI recipient with access to the adjustment of low and high frequency sound balance, known as Bass and Treble respectively. The clinical study is designed to evaluate the safety and effectiveness of recipient controlled Bass and Treble.

Subjects will have access to the Bass and Treble controls during a 4 week take-home period, and will complete questionnaires and diaries to provide descriptive data on the Bass and Treble adjustments made during take home use, and the success of these adjustments.

Pre and post intervention speech test results will be used to evaluate the effect of access to Bass and Treble controls on speech perception. The post intervention questionnaire will provide information on the overall ratings of the Bass and Treble controls.

ELIGIBILITY:
Inclusion Criteria:

1. Six years of age or older
2. At least 3 months experience with the CP810, CP910 or CP920 sound processor
3. At least 3 months experience with the CI24RE or CI500 series implant
4. Willingness to participate in and to comply with all requirements of the protocol

Exclusion Criteria:

1. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedure and prosthetic device
2. Additional disabilities that would prevent participation in evaluations

Ages: 6 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Non-inferior speech perception with preferred Bass and Treble settings compared to the baseline Bass and Treble settings | 8 weeks
  Co-primary endpoint #1: This endpoint is to test that speech perception scores in noise with preferred Bass and Treble settings are non-inferior to the baseline settings. Subjects will be tested at visit one with their own settings (Baseline), and then again after four weeks use of the Bass and Treble feature. The speech signal will arrive from zero degrees azimuth at a level of 65 dB SPL, the noise will also arrive from zero degrees azimuth, however the noise will adapt according to subject responses.
  o-primary endpoint #2: This endpoint is to test that speech perception scores in quiet with preferred Bass and Treble settings are non-inferior to the baseline settings. Subjects will be tested at visit one with their own settings (Baseline), and then again after four weeks use of the Bass and Treble feature. The speech signal will arrive from zero degrees azimuth at a level of 50 dB SPL.

SECONDARY OUTCOMES:
Non-inferior sentence recognition in four-talker babble noise with Bass and Treble values set to the minimum (-6 Bass, - 6 Treble) compared to the baseline condition when the speech and noise are from the front | 8 weeks
  Secondary endpoint #1: This endpoint is to test that speech perception scores in noise with Bass and Treble settings set to minimum (-6, -6) are non-inferior to the baseline settings. Subjects will be tested at visit one. The speech signal will arrive from zero degrees azimuth at a level of 65 dB SPL, the noise will also arrive from zero degrees azimuth, however the noise will adapt according to subject responses.

OTHER OUTCOMES:
Subjective daily diary data on the success of the daily Bass and Treble changes made during take-home use | 8 weeks
Questionnaire data on the overall subjective ratings of the Bass and Treble controls (importance, confidence, ease and satisfaction) | 8 weeks
Incidence of adverse events as well as the severity, relationship to treatment, outcome and actions taken will be listed for each subject and summarised. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chris D Warren, Audiology, Study Director — Employee
Locations (2):
- Australia (2):
  - Sydney Cochlear Implant Centre, Sydney, New South Wales
  - Cochlear Limited, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: No
Identifiable data will not be made available to the public. Data will be kept in a secure, locked environment and only the researchers working on the study, relevant authorities and authorised representatives will have access to it.
  Subject health records and any information obtained during the research project are subject to inspection (for the purpose of verifying the procedures and the data) by the Food and Drug Administration (FDA) of the United States of America, other national drug regulatory authorities and such as the Australian Government's Therapeutic Goods Administration (TGA), local Ethics Committees, and other duly authorised representatives of the Sponsor, or as required by law.
  Study subjects have consented to this.